CLINICAL TRIAL: NCT00099476
Title: Effects of Cocoa Consumption on Insulin Sensitivity and Capillary Recruitment in Subjects With Essential Hypertension
Brief Title: Effects of Dark Chocolate on Insulin Sensitivity in People With High Blood Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050047; 05-AT-0047
Record Dates: First submitted 2004-12-14; First posted 2004-12-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-16

CONDITIONS: Hypertension
Keywords: Epicatechin; Polyphenols; Chocolate; Insulin Resistance; Endothelial Dysfunction; Hypertension
MeSH Terms: conditions — Hypertension; Insulin Resistance

INTERVENTIONS:
Behavioral: Effects of dark chocolate

SUMMARY:
This study will examine whether dark chocolate affects the way patients with hypertension (high blood pressure) respond to insulin, a hormone secreted by the pancreas that regulates blood glucose (sugar) levels. In many people with hypertension, insulin is not as effective in helping the body use glucose. This is called insulin resistance. Insulin also increases blood flow into muscle by opening inactive blood vessels. Laboratory studies suggest that eating dark chocolate may improve blood pressure. This study will determine whether dark chocolate improves insulin resistance or changes how blood vessels react to insulin in hypertensive people.

People between 21 and 65 years of age who have high blood pressure and are not pregnant may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests.

Participants refrain from eating foods containing chocolate or cocoa for 1 week and then come to the clinic on three separate occasions 3 weeks apart for a glucose clamp test and contrast ultrasound, described below. At the first glucose clamp test, subjects are randomly assigned to drink either a cocoa drink with high anti-oxidant content or one with a very low content of anti-oxidant. Each drink will be taken twice a day for 2 weeks. At the end of the 2 weeks, they return for a second glucose clamp test. At the second test, they stop taking the cocoa drink for 1 week and then start again for another 2 weeks. For this 2-week period, those who were given the high anti-oxidant content cocoa drink the first 2 weeks will take the placebo, very low anti-oxidant drink this time, and those who took the placebo will now have the high anti-oxidant cocoa drink. After this 2 weeks of taking the cocoa drink or placebo, they then take the third and last glucose clamp test.

Glucose clamp test: This test measures how the body responds to insulin. Subjects fast the night before each test and do not eat until the test is over, usually in the early afternoon. For the test, the subject lies in a bed or reclines in a chair. A needle is placed in a vein in each arm - one for collecting blood samples and the other for infusing glucose, insulin, and a potassium solution. Blood glucose and insulin levels are measured frequently during the test and the rate of the glucose infusion is adjusted to keep blood glucose at the baseline (fasting) level. Blood samples are tested for blood count, electrolytes, liver function...

DETAILED DESCRIPTION:
Dark chocolate and other cocoa products contain antioxidants including the polyphenol epicatechin that have beneficial effects on vascular function. Oral consumption of dark chocolate lowers blood pressure in elderly subjects with isolated systolic hypertension while drinking cocoa acutely improves flow-mediated vasodilation in subjects with cardiovascular risk factors. Work from our lab and elsewhere has shown that regulation of hemodynamic and metabolic homeostasis are coupled such that subjects with essential hypertension are also insulin resistant. Therefore, we hypothesize that cocoa consumption will improve both blood pressure and insulin sensitivity in subjects with essential hypertension. To test this hypothesis, we will conduct a randomized double-blind, crossover study in subjects with essential hypertension to evaluate the effects of cocoa versus placebo on blood pressure, insulin sensitivity, and insulin-mediated capillary recruitment in skeletal muscle. After a 7 day cocoa-free run-in period, subjects will be randomized to receive 15 consecutive daily doses of either cocoa drink (150 ml twice a day with a total of 900 mg of polyphenols and 237 kcal) or polyphenol poor placebo drink (150 ml twice a day with a total of 36 mg of polyphenols and 234 kcal). After the 15 day treatment period, the subjects will enter a 1 week cocoa-free washout period followed by cross-over to the other treatment. Subjects will be counseled to maintain an isocaloric diet during the study. Blood pressure, insulin sensitivity, and insulin-mediated capillary recruitment will be assessed in each subject after the run-in period, after 15 days of treatment, and after completion of the cross-over. Blood pressure will also be measured every Monday, Wednesday, and Friday for the duration of the study. Insulin sensitivity will be measured using the hyperinsulinemic euglycemic glucose clamp technique. Insulin-stimulated capillary recruitment in forearm skeletal muscle will be measured by ultrasound with "microbubble" contrast during the glucose clamp studies. Peak and trough plasma epicatechin levels will be measured prior to each glucose clamp study using an HPLC assay. This study will determine if short-term oral administration of cocoa is effective at lowering blood pressure, improving insulin sensitivity, and restoring vascular function in subjects with essential hypertension. This is highly relevant to major public health problems such as diabetes, obesity, hypertension, and cardiovascular diseases where insulin resistance and vascular dysfunction are important pathophysiological components.

ELIGIBILITY:
* INCLUSION CRITERIA

Hypertensive subjects between the ages of 21 - 65 years in good general health except for mild to moderate hypertension (blood pressure between 140/95 and 170/110 off medication), on no medication or nutritional supplements except for antihypertensive agents, anti-cholesterol drugs or birth control agents. Subjects will be taken off all antihypertensive OTC supplements and anti-cholesterol drugs for one week prior to study and for the duration of the study. Women on birth control will remain on their regime. During the time subjects receive no antihypertensive therapy, their blood pressure will be monitored at least daily (either at home, in the clinic, or at another convenient facility). If a subject's blood pressure exceeds 170/110 on three determinations over a period of at least 15 minutes, the subject will be withdrawn from the study and appropriate antihypertensive therapy resumed. In addition, if the subject's blood pressure exceeds 160/100 during measurements on three consecutive days, the subject will be withdrawn from the study and appropriate antihypertensive therapy resumed.

EXCLUSION CRITERIA

Subjects will be excluded if they have diabetes, pregnancy, liver disease, pulmonary disease, renal insufficiency, coronary heart disease, heart failure, peripheral vascular disease, coagulopathy, actively smoked tobacco within last two years, in treatment for any form of cancer, positive tests for HIV, hepatitis B or C, or take systemic corticosteroids. These conditions are all known to adversely influence insulin sensitivity.

Subjects will be excluded if they have a history of malignant hypertension, aortic aneurysm or stroke.

Subjects with known hypersensitivity to octafluoropropane or with known cardiac shunts will also be excluded from participating because of potential adverse effects from microbubble contrast agent.

Subjects will be excluded if they are unable to give informed consent for all procedures.

Children are excluded from this study because children are not typically hypertensive.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2004-12-10; Study Completion 2009-04-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ferrannini E, Buzzigoli G, Bonadonna R, Giorico MA, Oleggini M, Graziadei L, Pedrinelli R, Brandi L, Bevilacqua S. Insulin resistance in essential hypertension. N Engl J Med. 1987 Aug 6;317(6):350-7. doi: 10.1056/NEJM198708063170605. PMID 3299096
- [Background] Modan M, Halkin H, Almog S, Lusky A, Eshkol A, Shefi M, Shitrit A, Fuchs Z. Hyperinsulinemia. A link between hypertension obesity and glucose intolerance. J Clin Invest. 1985 Mar;75(3):809-17. doi: 10.1172/JCI111776. PMID 3884667
- [Background] Zavaroni I, Mazza S, Dall'Aglio E, Gasparini P, Passeri M, Reaven GM. Prevalence of hyperinsulinaemia in patients with high blood pressure. J Intern Med. 1992 Mar;231(3):235-40. doi: 10.1111/j.1365-2796.1992.tb00529.x. PMID 1556520
- [Derived] Muniyappa R, Hall G, Kolodziej TL, Karne RJ, Crandon SK, Quon MJ. Cocoa consumption for 2 wk enhances insulin-mediated vasodilatation without improving blood pressure or insulin resistance in essential hypertension. Am J Clin Nutr. 2008 Dec;88(6):1685-96. doi: 10.3945/ajcn.2008.26457. PMID 19064532